CLINICAL TRIAL: NCT06469710
Title: A Trial to Evaluate the Effect of Applying Leukapheresis to Enrich CTCs in Patients With Metastatic Prostate Cancer
Brief Title: A Trial to Evaluate the Effect of Applying Leukapheresis to Enrich CTCs in mPCa Patients
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Liang Dong, vice president of Renji Hospital, RenJi Hospital
Other Study IDs: LY2024-076-A
Record Dates: First submitted 2024-06-13; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer; Circulating Tumor Cell; Leukapheresis
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating | interventions — Leukapheresis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: leukapheresis — Leukapheresis employs the density differential between leukocytes and other blood components to selectively separate leukocytes and return all other components of the blood to the patient. It can process multiple blood volumes in the body circulation, thereby enabling the concentration of nucleated cells to be significantly increased. The procedure is performed while maintaining no significant change in the patient's circulating blood volume, and it is a routine clinical procedure that is well tolerated and safe. CTC can be greatly enriched in a concentrated sample of leukocytes because it has a similar density to that of leukocytes and other nucleated cells. The density of CTCs is similar to that of nucleated cells, such as leukocytes, which enables their enrichment in single leukocyte concentrate samples.

SUMMARY:
The goal of this observational study is to compare the number of CTCs enriched by both sampling methods, leukapheresis and collection of peripheral blood in metastatic prostate cancer patients. The main questions it aims to answer are:

1. The advantages and disadvantages of two sampling methods for further diagnosis and treatment;
2. How to obtain further information on the tumour biology of CTC;
3. The mechanisms of prostate cancer invasion and metastasis Participants will have 7.5mL of peripheral blood taken as well as undergo leukapheresis.

ELIGIBILITY:
Inclusion Criteria:

1. male, aged 18-75 years; and
2. Evidence of metastasis (positive finding of metastasis on one of the following tests: CT and MRI; whole-body nuclear bone imaging, fluoride PET and PET-CT, cholinergic PET-CT and MRI; prostate-specific membrane antigen-targeted PET-CT); or clinical diagnosis of metastatic prostate cancer (tumour stage of T3 and above) by pathology of aspiration/surgical biopsy;
3. Good general condition, ECOG score 0-1, able to tolerate leukapheresis;
4. Normal haematological analysis, liver and renal function tests at screening;
5. Subjects (or their legal representatives) can understand the informed consent form.

Exclusion Criteria:

1. those who have received systemic combination therapy for tumours within 5 years;
2. those with poor general condition, severe haemodynamic instability, malignant arrhythmias, cachexia and infections
3. those with coagulation disorders, DIC or reduced platelets;
4. those receiving exogenous plasma at the time of the trial;

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic prostate cancer with the following specific subject recruitment criteria:
  1. Clinical diagnosis of metastatic prostate cancer with tumour stage of T3 or above;
  2. Metastatic signs on relevant imaging tests, including CT and MRI, whole-body nuclear bone imaging, fluoride PET and PET-CT, cholinergic PET-CT and MRI, and prostate specific membrane antigen (PSMA)-targeted PET-CT;
  3. After radical prostatectomy for prostate cancer with indication of biochemical recurrence (PSA>0.2ng/mL);
  4. Those with metastatic prostate cancer diagnosed by puncture or postoperative pathology;
  5. Previous medical history and treatment history.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-25 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of circulating tumor cells | The leukapheresis takes about 2 hours, and CTCs number will be measured in 24 hours after sampling.
  Measurement of the number of CTCs enriched from different samples

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, Shanghai, China